CLINICAL TRIAL: NCT02036333
Title: The Role of Cerebral Oximetry in Pediatric Concussion Assessment
Status: Terminated | Type: Observational
Why Stopped: Key Personnel Left Institution Prior to Study Completion
Sponsor: Johns Hopkins University (Other)
Collaborators: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: NA_00078909
Record Dates: First submitted 2014-01-13; First posted 2014-01-15 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Concussion, Brain; Concussion, Mild; Traumatic Brain Injury
Keywords: near infrared spectroscopy; pediatrics
MeSH Terms: conditions — Brain Concussion; Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Concussion Group
- Control Group

SUMMARY:
The purpose of this study is to determine whether there is a difference in cerebral oxygenation as measured by near-infrared spectroscopy (NIRS) in children with concussion and healthy controls.

ELIGIBILITY:
INCLUSION CRITERIA:

All Participants

* Age 10-18 years at time of visit

Concussion Group

* Present to JHH PED within the first 24 hours following trauma.
* Diagnosis of concussion as defined by the 3rd International Conference on Concussion in Sport (McCrory), including the presence of any one or more of the following:

  1. Symptoms (ie. headache, neck pain, nausea/vomiting, dizziness, blurred vision, balance problems, sensitive to light, sensitivity to noise, feeling slowed down, feeling in a fog, difficulty concentrating, difficulty remembering, fatigue, confusion, drowsiness, more emotional, irritability, sadness, nervous)
  2. Physical Signs (ie. loss of consciousness, unsteadiness)
  3. Impaired brain function (ie. confusion)
* Glasgow Coma Score of 13-15 upon arrival to JHH PED.
* Loss of consciousness of less than 15 minutes (if applicable).
* No structural intracranial injuries identified on neuroimaging (if completed).

EXCLUSION CRITERIA

All Participants

* History of prior concussion or traumatic brain injury within preceding 6 weeks.
* History of prior intracranial disease or mass (ie. tumor, intraventricular hemorrhage, etc.)
* Presence of intracranial hardware.
* Complaints of respiratory distress, tachypnea or hypoxia, which may affect regional cerebral oxygen saturation.
* Inability to stand secondary to lower extremity disease or trauma, which is required for completion of SCAT2.
* Inability to complete SCAT2 questionnaire secondary to developmental delay.
* Child in foster care or legal guardian not available.
* Participant known to be pregnant, which alters total body blood flow and likely affects regional cerebral oxygen saturation.
* Non-English speaking.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: This pilot study will employ a prospective cohort study design. Children aged 10-18 years will be recruited within the Johns Hopkins Hospital Pediatric Emergency Department (JHH PED) to participate in this study. All children must be conversant in English.
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2015-06-30 (Actual); Study Completion 2015-06-30 (Actual)

PRIMARY OUTCOMES:
Difference in mean baseline regional cerebral oxygen saturation as measured by near-infrared spectroscopy between children with mild traumatic brain injury and controls. | At presentation (Day 0)

SECONDARY OUTCOMES:
Difference in the change in regional cerebral oxygen saturation during handgrip exercise between children with mild traumatic brain injury and controls. | At presentation (Day 0)
Difference in Sport Concussion Assessment Tool 2 (SCAT2) total score between patients with mild traumatic brain injury and controls. | At presentation (Day 0)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Anders, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University Pediatric Emergency Medicine, Baltimore, Maryland, United States